CLINICAL TRIAL: NCT05036135
Title: IMPAHCT: A Phase 2b/3, Randomized, Double-Blind, Placebo-Controlled, 24-Week Dose Ranging and Confirmatory Study to Evaluate the Safety and Efficacy of AV-101 in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: A Study of AV-101 (Dry Powder Inhaled Imatinib) in Patients With Pulmonary Arterial Hypertension (PAH)
Acronym: IMPAHCT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The IMPAHCT study demonstrated that while inhaled imatinib was well tolerated, it did not prove to be efficacious at any of the doses of AV-101 evaluated in the study.
Sponsor: Aerovate Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AV-101-002
Record Dates: First submitted 2021-08-16; First posted 2021-09-05 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary Arterial Hypertension; Lungs; Pulmonary; PAH; AV-101; imatinib; IMPAHCT
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- AV-101 10 mg (Experimental)
  Interventions: Drug: AV-101
- AV-101 35 mg (Experimental)
  Interventions: Drug: AV-101
- AV-101 70 mg (Experimental)
  Interventions: Drug: AV-101
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AV-101 — AV-101 (imatinib) administered via dry powder inhalation
  Arms: AV-101 10 mg; AV-101 35 mg; AV-101 70 mg
Drug: Placebo — Placebo administered via dry powder inhalation
  Arms: Placebo

SUMMARY:
IMPAHCT: Inhaled iMatinib Pulmonary Arterial Hypertension Clinical Trial is a Phase 2b/Phase 3 study to evaluate the safety and efficacy of AV-101 (dry powder inhaled imatinib) in patients with Pulmonary Arterial Hypertension (PAH). The Phase 2b part of the study will assess three doses to establish an optimal dose for the Phase 3 part of the study. The Phase 2b primary endpoint will be the placebo corrected change in pulmonary vascular resistance (PVR). The Phase 3 primary endpoint will be the placebo corrected change in 6-minute walk distance (6MWD) after 24 weeks of treatment.

ELIGIBILITY:
Key Inclusion Criteria

* PAH belonging to one of the subgroups:

  1. I/HPAH, PAH-CTD,
  2. PAH due to drugs and/or toxins/chemicals (having been in the care of the investigator for at least one year with no relapses of drug or toxin/chemical abuse),
  3. HIV associated or
  4. PAH due to repaired congenital heart disease (at least 1 year since repair)
* World Health Organization (WHO) Functional Class II, III or IV symptoms
* Stable concomitant background therapy of at least one PAH approved medications
* Able to walk a distance of at least 100 m but no more than 475 m during the Screening 6-minute walk tests.

Key Exclusion Criteria

* Pulmonary hypertension (PH) belonging to Groups 2 to 5
* A history of left-sided heart disease
* Pregnant or breast-feeding females

Additional criteria may apply, per protocol

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2024-08-09 (Actual); Study Completion 2024-08-09 (Actual)

PRIMARY OUTCOMES:
Phase 2b: Change from Baseline in Pulmonary Vascular Resistance (PVR) | 24 weeks
Phase 3: Change from Baseline in Six Minute Walk Distance (6MWD) | 24 weeks

SECONDARY OUTCOMES:
Phase 2b: Change from Baseline in N-terminal pro B-type natriuretic peptide (NT-proBNP) | 24 weeks
Phase 2b: Change from Baseline in Six Minute Walk Distance (6MWD) | 24 weeks
Phase 2b: Time to Clinical Worsening | 24 weeks
Phase 2b: Proportion of Subjects with Improvement in WHO Functional Class | 24 weeks
Phase 2b: Change from Baseline in Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) Lite 2.0 Risk Score | 24 weeks
  REVEAL Lite 2.0 risk scores range from 1 to 14; a higher score represents higher risk
Phase 2b: Change from Baseline in Health-Related Quality of Life emPHasis-10 Questionnaire Score | 24 weeks
  emPHasis-10 questionnaire scores range from 0 - 50; a higher score represents a higher symptom burden
Phase 3: Change from Baseline in NT-proBNP | 24 weeks
Phase 3: Time to Clinical Worsening | 24 weeks
Phase 3: Proportion of Subjects with Improvement in WHO Functional Class | 24 weeks
Phase 3: Change from Baseline in Registry to Evaluate Early and Long-Term PAH Disease Management (REVEAL) Lite 2.0 Risk Score | 24 weeks
  REVEAL Lite 2.0 risk scores range from 1 to 14; a higher score represents higher risk
Phase 3: Change from Baseline in Pulmonary Arterial Hypertension-Symptoms and Impact (PAH-SYMPACT) Questionnaire Score | 24 weeks
  PAH-SYMPACT is a patient reported outcome instrument developed to assess PAH symptoms and impacts

CONTACTS AND LOCATIONS:
Locations (128):
- United States (39):
  - Arizona Pulmonary Specialists, Ltd., Phoenix, Arizona
  - University of Arizona, Department of Medicine, Tucson, Arizona
  - UCLA/David Geffen School of Medicine-Pulmonary and Criticial Care, Los Angeles, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Pulmonary & Critical Care, Los Angeles, California
  - Dept of Veterans Affairs Greater Los Angeles Healthcare System, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of California, San Francisco, California
  - LA Biomedical Research Institute Harbor, Torrance, California
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - George Washington University Medical Faculty Associates, Inc., Washington D.C., District of Columbia
  - Mayo Clinic Florida, Jacksonville, Florida
  - Orlando Heart Center, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University Health, Indianapolis, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tufts Medical Center, Inc., Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center- Hematology/Oncology Section, Omaha, Nebraska
  - The Unviersity of New Mexico - UNM Hospitals, Albuquerque, New Mexico
  - New York-Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York
  - NYU Langone Seaport, New York, New York
  - Duke University Medical Center - Duke South Clinic, Durham, North Carolina
  - The Lindner Center for Research and Education, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Bend Memorial Clinic, Oregon City, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Stat Care Pulmonary Consultants, PLLC, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Sentara Medical Group - Sentara Pulmonary & Critical Care Specialists, Norfolk, Virginia
- Argentina (7):
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Nexo Salud Investigación Clínica, Buenos Aires
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Cardiología Palermo, CABA
  - Insituto Medico DAMIC, Córdoba
  - Hospital Italiano de Cordoba, Córdoba
  - Hospital Dr. Jose Maria Cullen, Santa Fe
- Australia (9):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord West, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - The Prince Charles Hospital, Chermside, Queensland
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Adelaide Hospital, Adelaide
  - Fiona Stanley Hospital, Murdoch
- AKH - Medizinische Universitat Wien, Vienna, Austria
- Belgium (2):
  - Hopital Erasme - Cliniques Universitaires de Bruxelles, Brussels
  - UZ Leuven, Leuven
- Brazil (2):
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Heart Institute - University of Sao Paulo, São Paulo
- Canada (4):
  - The Governors of the University of Calgary, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - London Health Science Centre, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Centro de Investigaciones Clinicas de la Universidad Catolica, Santiago, Chile
- China (9):
  - Peking Union Medical College Hospital, Beijing
  - Chongqing Medical University - The First Affiliated Hospital, Chongqing
  - Guangdong Provincial People's Hospital, Guangdong
  - Central South University - The Second Xiangya Hospital, Hunan
  - Yanan Hospital of Kunming City, Kunming
  - Gansu Provincial People's Hospital, Lanzhou
  - Southeast University (SEU) - Zhongda Hospital, Nanjing
  - Shanghai Pulmonary Hospital, Shanghai
  - Tianjin Medical University General Hospital, Tianjin
- Vseobecna fakultni nemocnice v Praze, Prague, Czechia
- France (5):
  - Groupement Hospitalier Sud - Hôpital Bicêtre, Le Kremlin-Bicêtre, Cedex
  - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron
  - Hôpital Nord - CHU Marseille, Marseille
  - Hopital Arnaud de Villeneuve, Montpellier
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (4):
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giesen
  - Universitaetsklinikum Heidelberg, Heidelberg
  - München Klinik Bogenhausen, München
- Greece (3):
  - University General Hospital Attikon, Athens
  - Cardiosurgery Hospital, Kallithea
  - AHEPA General Hospital of Thessaloniki, Thessaloniki
- Israel (3):
  - The Lady Davis Carmel Medical Center, Haifa
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti - Foggia, Foggia
  - Ospedale San Giuseppe - Fatebenefratelli, Milan
  - Azienda Socio Sanitaria Territoriale di Monza, Monza
  - Azienda Ospedaliera Vincenzo Monaldi, Napoli
  - Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Azienda Ospedaliera Universitaria Policlinico Umberto I, Rome
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Mexico (4):
  - CICUM San Miguel, Guadalajara, Jalisco
  - Unidad de Investigacion Clinica en Medicina S.C., Monterrey, Nuevo León
  - Instituto Nacional de Cardiologia Dr Ignacio Chavez Rivera, Mexico City
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario, Monterrey
- Amsterdam UMC, Locatie VUMC, Amsterdam, Netherlands
- Poland (4):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Bieganski Provincial Specialist Hospital, Lodz
  - Szpital Kliniczny Przemienienia Pańskiego UM im. Marcinkowskiego, Poznan
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego, Wroclaw
- Portugal (3):
  - Hospital Garcia de Orta, EPE, Almada
  - Hospital Pulido Valente, Lisbon
  - CHUPorto, Porto
- Cardiopulmonary Research Center, Guaynabo, Puerto Rico
- Singapore (2):
  - National University Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Center of Chest Disease Johannesburg, Johannesburg, South Africa
- Spain (9):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hosp. Universitario Gran Canaria Doctor Negrin, Las Palmas de Gran Canaria
  - Hospital 12 de Octubre, Madrid
  - Universidad Autonoma de Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital universtario de Salamanca, Salamanca
  - Hosp. Universitario Marques de Valdecilla, Santander
  - Hospital Universitario de Toledo, Toledo
- Norrlands Universitetssjukhus, Umeå, Sweden
- United Kingdom (4):
  - Imperial College Healthcare NHS Trust, London, England
  - Golden Jubilee National Hospital, Glasgow
  - Royal Brompton Hospital, London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gillies H, Chakinala MM, Dake BT, Feldman JP, Hoeper MM, Humbert M, Jing ZC, Langley J, McLaughlin VV, Niven RW, Rosenkranz S, Zhang X, Hill NS. IMPAHCT: A randomized phase 2b/3 study of inhaled imatinib for pulmonary arterial hypertension. Pulm Circ. 2024 Mar 25;14(1):e12352. doi: 10.1002/pul2.12352. eCollection 2024 Jan. PMID 38532768
- [Derived] Gillies H, Niven R, Dake BT, Chakinala MM, Feldman JP, Hill NS, Hoeper MM, Humbert M, McLaughlin VV, Kankam M. AV-101, a novel inhaled dry-powder formulation of imatinib, in healthy adult participants: a phase 1 single and multiple ascending dose study. ERJ Open Res. 2023 Mar 13;9(2):00433-2022. doi: 10.1183/23120541.00433-2022. eCollection 2023 Mar. PMID 36923571